CLINICAL TRIAL: NCT02193932
Title: EEG-triggered fMRI in Epilepsy Patients
Brief Title: Electroencephalogram (EEG) Triggered Functional Magnetic Resonance Imaging (fMRI) in Epilepsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-100
Record Dates: First submitted 2014-07-10; First posted 2014-07-18 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
Keywords: EEG triggered; fMRI; epilepsy; intractable
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EEG Triggered fMRI using Micro Maglink (Experimental): EEG Triggered fMRI to be performed using the Micro Maglink
  Interventions: Other: EEG Triggered fMRI using Micro Maglink

INTERVENTIONS:
Other: EEG Triggered fMRI using Micro Maglink

SUMMARY:
A prospective exploratory study in patients with drug resistant epilepsy with a target comparison of long term outcome. NeuroScan software modules and a MagLink will be used to acquire EEG in combination with MRI/fMRI data. The MagLink system is used for obtaining integrated EEG and Event Related Potential (ERP) recordings while the subject is inside the MRI machine, without compromising the raw EEG data.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory epilepsy cases, referred by the service of Neurology. These are cases whose pathophysiology is resistant to treatment, including change in medication and or added medication.
2. Patients will be included if they agree to sign an Institutional Review Board approved written consent.

Exclusion Criteria:

1. Patients with overt symptoms or signs of anxiety than cannot cooperate during the recording inside the scanner, unless consent is given for the procedure to be performed with sedation by the anesthesia department.
2. Patients who meet the regular exclusion criteria for Magnetic Resonance Imaging (MRI) studies per the prescreening form reviewed with all patients prior to exams

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with at least 40 interictal epileptic discharges during the fMRI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Gonzalez-Arias, MD, Principal Investigator — Baptist Health South Florida
Locations (1):
- Baptist Hospital, Miami, Florida, United States